CLINICAL TRIAL: NCT02075918
Title: Integrated Approaches for Identifying Molecular Targets in Alcoholic Hepatitis
Acronym: InTeam
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of Wisconsin, Madison (Other); King's College London (Other); Veterans Medical Research Foundation (Other); Hospital Vall d'Hebron (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Yale University (Other); Columbia University (Other); Weill Medical College of Cornell University (Other); University of Alberta (Other); TecSalud Investigación Clínica (Other)
Responsible Party: Principal Investigator, Ramon Bataller, Professor, University of Pittsburgh
Other Study IDs: 12-2016; 1U01AA021908-01 (NIH)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Alcoholic Hepatitis; Control Patients
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Whole Blood DNA, PBMCs, Urine, Stool, Liver Biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: To improve the diagnosis and assessment of severity of acute alcoholic hepatitis Participants: Patients admitted to one of ten centers with acute alcoholic hepatitis Procedures (methods): Consecutive patients admitted with acute alcoholic hepatitis will be enrolled in an NIH U01 study of acute alcoholic hepatitis where liver tissue, blood and stool will be collected to discover and validate factors associated with diagnosis, severity of disease and survival.

DETAILED DESCRIPTION:
The development of new targeted therapies for alcoholic hepatitis (AH) is one of the more urgent needs in clinical hepatology. To reach this goal, large multidisciplinary networks are required. The proposed initiative "Integrated Approaches for Identifying Molecular Targets in Alcoholic Hepatitis" (InTeam) will coordinate a multidisciplinary group composed of clinicians, physician-scientists, basic scientists and bioinformatics experts. The overarching hypothesis of InTeam is that the most rational way to provide a useful framework for future clinical trials in (AH) consists of the (i) determination of key drivers of the disease process, (ii) classification of molecular profiles and subtypes of AH, and (iii) identification of "druggable" targets based on both key drivers and molecular classification. Moreover, mouse models for AH are lacking making it impossible to evaluate promising targets in preclinical mouse studies in a meaningful manner. For this purpose, InTeam will integrate data obtained from molecular pathology studies in human AH and functional studies of key pathways in animal models. The proposed InTeam consortium includes three research projects, ten clinical centers, a Human Biorepository and a Mouse Models Core. The Human Biorepository Core will generate the to-date largest collection of samples from patients with AH from 10 academic liver centers and a comprehensive database that will serve as a basis for the proposed translational studies and be a valuable asset for the broader scientific community. The Mouse Models core will conduct murine studies after establishing and evaluating mouse models of AH based on the pathophysiology and molecular drivers of human AH determined by this consortium.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 ≥ and ≤ 70 years of age.
* Active alcohol abuse within the past 3 months.
* Has an Aspartate Aminotransferase (AST) > Alanine Aminotransferase (ALT).
* Elevated Total Bilirubin level > 3.0.
* Absence of autoimmune liver disease (ANA>1/320).
* Absence of hepatitis B infection.
* A liver biopsy, and/or a clinical picture consistent with alcoholic hepatitis.
* The "Start Date" (is the date of the liver biopsy or ≤ to 1 week [72 hours is preferred] from the time of admission).

Exclusion Criteria:

* Hepatocellular carcinoma.
* Complete portal vein thrombosis.
* Advanced or terminal extrahepatic diseases.
* Lack of consent to participate in the study.
* Pregnancy.
* Received more than 3 days of treatment with (prednisolone or pentoxifyllin) prior to start date.

Control patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an episode of alcoholic hepatitis fulfilling the inclusion criteria will be eligible to participate in the study. Those patients who meet one or more exclusion criteria will not be included.
  Control patients
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2014-05; Primary Completion 2019-05 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis and Severity of Alcoholic Hepatitis | 3 months after end of Study
  Utilizing liver tissue, blood samples, and stool and urine samples, InTeam will aim to discover and validate factors associated with the diagnosis and severity of Alcoholic hepatitis.

SECONDARY OUTCOMES:
Major Liver Complications | 3 months after end of study
  As an observational study, we will collect data regarding major liver complications such as, ascites, renal failure, encephalopathy, and bleeding.
Death/Transplantation | 3 months after end of study
  As an observational study, we will collect the data regarding number the survival of Alcoholic Hepatitis by considering deaths and transplantations.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Bataller, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lang S, Duan Y, Liu J, Torralba MG, Kuelbs C, Ventura-Cots M, Abraldes JG, Bosques-Padilla F, Verna EC, Brown RS Jr, Vargas V, Altamirano J, Caballeria J, Shawcross D, Lucey MR, Louvet A, Mathurin P, Garcia-Tsao G, Ho SB, Tu XM, Bataller R, Starkel P, Fouts DE, Schnabl B. Intestinal Fungal Dysbiosis and Systemic Immune Response to Fungi in Patients With Alcoholic Hepatitis. Hepatology. 2020 Feb;71(2):522-538. doi: 10.1002/hep.30832. Epub 2019 Aug 20. PMID 31228214